CLINICAL TRIAL: NCT03074500
Title: A Randomized Controlled Trial Comparing the Effects of Kinesiology Taping With Exercise, Sham Taping With Exercise and Exercise Alone for Lateral Epicondylitis
Brief Title: Kinesiotaping in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.2017.004
Record Dates: First submitted 2017-03-01; First posted 2017-03-08 (Actual); Results first posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Lateral Epicondylitis
Keywords: Kinesio taping; lateral epicondylitis; tennis elbow; treatment
MeSH Terms: conditions — Tennis Elbow | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: To ensure group concealment, randomization will be done by using opaque, sealed envelopes which the assessors will be blinded to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Kinesiotaping (Experimental): Kinesio taping by using space correction and fascia correction techniques every 3 days for 2 weeks in addition to exercises
  Interventions: Device: Kinesiotaping; Other: Exercise
- Sham taping (Sham Comparator): Sham taping without using any techniques every 3 days for 2 weeks in addition to exercises
  Interventions: Other: Sham taping; Other: Exercise
- Control (Other): Stretching and strengthening exercises of wrist
  Interventions: Other: Exercise

INTERVENTIONS:
Device: Kinesiotaping — Kinesio tape will be applied by using space correction and fascia correction technique on forearm of the patients for the treatment of lateral epicondylitis
  Arms: Kinesiotaping
Other: Sham taping — Sham taping will be performed without using any technique
  Arms: Sham taping
Other: Exercise — Stretching exercises of wrist 30 seconds to one minute, twice a day and strengthening exercises will performed be 10 repetitions in 2 or 3 series. .

SUMMARY:
The aim of this study is to compare the effects of kinesiology taping with exercise, sham taping with exercise and exercise alone for lateral epicondylitis.

DETAILED DESCRIPTION:
Lateral epicondylitis or tennis elbow is a often-encountered disorder of elbow which is characterized by tenderness and pain over lateral epicondylitis of humerus and grip weakness. The annual incidence of lateral epicondylitis has been reported to be %1-3 in general population. Lateral epicondylitis is commonly associated with repetitive overuse of wrist, activities including strong grip which in turn cause microtears and degenerative changes over the common origin of wrist and finger extensors on lateral epicondyle. New researches have shown that the underlying mechanism is degenerative rather than inflammatory. It has been proposed that the cause of pain may be mechanical discontinuity of collagen fibers or biochemical irritation that results from damaged tendon tissue that activates nociceptors. It has been suggested that eccentric loading has been shown to assist with tendon rehabilitation by improving collagen alignment and stimulating collagen cross-linkage formation, both of which can improve tensile strength.

Kinesio taping (KT) which is a new application of adhesive taping was designed by Kenzo Kase to avoid unwanted effects of conventional taping such as restricting range of motion (ROM) and limiting functional activities. The recommended tape application methods are outlined in 'Clinical Therapeutic Applications of the Kinesio Taping Method' 8. Elastic therapeutic tape has been designed to allow for a longitudinal stretch of up to 140% of its resting length and has been designed to approximate the elastic qualities of the human skin. In particular, the application of the tape over stretched muscle to create convolutions in the skin has been hypothesized to reduce pressure in the mechanoreceptors below the dermis, thereby decreasing nociceptive stimuli. Another mechanism which is claimed by the proponent of the tape is that convolutions are raised ridges of the tape and the skin that are thought to decompress underlying structures and allow for enhanced circulation by increased subcutaneous space. In the last few years, the use of KT has become increasingly popular in rehabilitation programs as an adjunct in the treatment. However, scientific evidence about its effect is insufficient.

The aim of this study is to compare the effects of kinesiology taping with exercise, sham taping with exercise and exercise alone for lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

1. Having had symptoms less than 12 weeks
2. Tenderness and pain over lateral epicondylitis
3. Provocation of the lateral elbow pain with at least one of the following tests - resisted middle finger extension (Maudley's test), resisted wrist extension or passive stretch of wrist extensors (Mill's test).

Exclusion Criteria:

1. Cervical spondylosis or radiculopathy
2. Diabetes mellitus
3. Neuropathy
4. Arthritis in the upper extremities
5. History of injection and physical therapy for lateral epicondylitis within the last three months
6. Pregnancy
7. History of surgery or acute trauma in the elbow
8. Allergy to tape

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gulseren Derya Akyuz, MD,Prof, Study Director — Marmara University School of Medicine, PM&R Department; Esra Giray, Principal Investigator — Marmara University School of Medicine, PM&R Department
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wegener RL, Brown T, O'Brien L. A randomized controlled trial of comparative effectiveness of elastic therapeutic tape, sham tape or eccentric exercises alone for lateral elbow tendinosis. Hand Therapy 2016;21(4):131-9.
- [Background] Kase K. Clinical therapeutic applications of the Kinesio taping methods. 2016.
- [Result] Lee SS, Kang S, Park NK, Lee CW, Song HS, Sohn MK, Cho KH, Kim JH. Effectiveness of initial extracorporeal shock wave therapy on the newly diagnosed lateral or medial epicondylitis. Ann Rehabil Med. 2012 Oct;36(5):681-7. doi: 10.5535/arm.2012.36.5.681. Epub 2012 Oct 31. PMID 23185733
- [Result] Kucuksen S, Yilmaz H, Salli A, Ugurlu H. Muscle energy technique versus corticosteroid injection for management of chronic lateral epicondylitis: randomized controlled trial with 1-year follow-up. Arch Phys Med Rehabil. 2013 Nov;94(11):2068-74. doi: 10.1016/j.apmr.2013.05.022. Epub 2013 Jun 22. PMID 23796685
- [Result] Struijs PA, Smidt N, Arola H, Dijk vC, Buchbinder R, Assendelft WJ. Orthotic devices for the treatment of tennis elbow. Cochrane Database Syst Rev. 2002;(1):CD001821. doi: 10.1002/14651858.CD001821. PMID 11869609
- [Result] Guo YH, Kuan TS, Chen KL, Lien WC, Hsieh PC, Hsieh IC, Chiu SH, Lin YC. Comparison Between Steroid and 2 Different Sites of Botulinum Toxin Injection in the Treatment of Lateral Epicondylalgia: A Randomized, Double-Blind, Active Drug-Controlled Pilot Study. Arch Phys Med Rehabil. 2017 Jan;98(1):36-42. doi: 10.1016/j.apmr.2016.08.475. Epub 2016 Sep 22. PMID 27666156
- [Result] Altan L, Kanat E. Conservative treatment of lateral epicondylitis: comparison of two different orthotic devices. Clin Rheumatol. 2008 Aug;27(8):1015-9. doi: 10.1007/s10067-008-0862-8. Epub 2008 Mar 26. PMID 18365136
- [Result] Dilek B, Batmaz I, Sariyildiz MA, Sahin E, Ilter L, Gulbahar S, Cevik R, Nas K. Kinesio taping in patients with lateral epicondylitis. J Back Musculoskelet Rehabil. 2016 Nov 21;29(4):853-858. doi: 10.3233/BMR-160701. PMID 27232082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was March 2017-May 2017 Setting: A university hospital outpatient clinics
Pre-assignment Details: Number of patients assessed for eligibility was 41. Among them,8 participants were excluded due to being inappropiate for the inclusion criteria (2 had concomittant radiculopathy, 2 were diagnosed as cubital tunnel syndrome, 2 were diagnosed as carpal tunnel syndrome and 2 of them had duration of symptoms were more than 12 weeks)
Groups:
- Kinesiotaping: Kinesio taping by using space correction and fascia correction techniques every 3 days for 2 weeks in addition to exercises
  Kinesio taping: Kinesio tape will be applied by using space correction and fascia correction technique on forearm of the patients for the treatment of lateral epicondylitis
  Exercise: Stretching exercises of wrist 30 seconds to one minute, twice a day and strengthening exercises will performed be 10 repetitions in 2 or 3 series. .
Period: Overall Study
Arm/Group | Kinesiotaping | Control | Sham Taping
Started | 11 | 11 | 11
Completed | 10 | 10 | 10
Not Completed | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Kinesiotaping: Kinesio taping by using space and fascia correction techniques on forearm of the patients for lateral epicondylitis treatment will be applied every 3 days for 2 weeks in addition to exercises.
  Exercise: Stretching exercises of wrist 30 seconds to one minute, twice a day and strengthening exercises will performed be 10 repetitions in 2 or 3 series.
- Sham Taping: Sham taping without using any techniques every 3 days for 2 weeks in addition to exercises
  Exercise: Stretching exercises of wrist 30 seconds to one minute, twice a day and strengthening exercises will performed be 10 repetitions in 2 or 3 series.
- Control: Only-exercises group: Stretching and strengthening exercises of wrist
  Exercise: Stretching exercises of wrist 30 seconds to one minute, twice a day and strengthening exercises will performed be 10 repetitions in 2 or 3 series.
- Total: Total of all reporting groups
Arm/Group | Kinesiotaping | Sham Taping | Control | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46.5 [32.5 to 53.5] | 45 [41.5 to 52.25] | 41.5 [34.75 to 53.25] | 45 [36.5 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 9 | 26
  Male | 1 | 2 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 10 | 30
Region of Enrollment [Number; unit: participants]
  Turkey | 10 | 10 | 10 | 30
Duration of Symptoms [Median (Inter-Quartile Range); unit: weeks] | 7 [5.5 to 8] | 8 [4 to 10.5] | 7 [5.5 to 12] | 8 [4 to 10]
Nirschl Score [Median (Full Range); unit: Scores on a scale] — Nirschl Scoring is a Likert scale ranging from 1 to 7 and classifying LE by the pain phase as a guide to the severity of the problem. Phase 1: Mild pain with exercise, resolves in 24 hours; Phase 2: Pain with exercise, exceeds 48 hours; Phase 3: Pain with exercise, does not alter activity; Phase 4: Pain with exercise, alters activity; Phase 5: Pain with heavy activities of daily living; Phase 6: Pain with light activities of daily living, intermitten pain at rest; Phase 7: Constant pain at rest, disrupts sleep.
  Scores on a scale | 5 [3 to 7] | 4.5 [3 to 5] | 5 [1 to 6] | 5 [1 to 7]
PRTEE (Patient rated tennis elbow evaluation) [Median (Inter-Quartile Range); unit: units on a scale] — PRTEE is a 15-item questionnaire designed tomeasure the forearm pain and disability in patients with LET. PRTEE allows patients to rate their levels of elbow pain and disability from 0 to 10 and consists of 2 subscales: 1) Pain subscale [5 items] (0 = no pain, 10 = worst imaginable) 2) Function subscale [Specific activities - 6 items, Usual activities - 4 items] (0 = no difficulty, 10 = unable to do). A total score can be computed on a scale of 100 (0 = no disability).
  units on a scale | 49 [43.88 to 73] | 53.75 [48.62 to 63] | 49.25 [41 to 57.5] | 51 [44.25 to 60.62]

OUTCOME MEASURES:

1. Primary Outcome: Patient Rated Tennis Elbow Evaluation (PRTEE)
Description: PRTEE is a 15-item questionnaire designed to measure the forearm pain and disability in patients with LE. PRTEE allows patients to rate their levels of elbow pain and disability from 0 to 10. Test consists of 2 subscales: 1) Pain subscale [5 items] (0 = no pain, 10 = worst imaginable) 2) Function subscale [Specific activities - 6 items, Usual activities - 4 items] (0 = no difficulty, 10 = unable to do). A total score can be computed on a scale of 100 (0 = no disability).
Time Frame: 0. week (Baseline), 2. week (After Treatment), 6. week (4 weeks After Treatment)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Kinesiotaping: Kinesio taping by using space correction and fascia correction techniques every 3 days for 2 weeks in addition to exercises
  Kinesio taping: Kinesio tape will be applied by using space correction and fascia correction technique on forearm of the patients for the treatment of lateral epicondylitis
  Exercise: Stretching exercises of wrist 30 seconds to one minute, twice a day and strengthening exercises will performed be 10 repetitions in 2 or 3 series.
- Sham Taping: Sham taping without using any techniques every 3 days for 2 weeks in addition to exercises
  Sham taping: Sham taping will be performed without using any technique
  Exercise: Stretching exercises of wrist 30 seconds to one minute, twice a day and strengthening exercises will performed be 10 repetitions in 2 or 3 series.
Arm/Group | Kinesiotaping | Sham Taping | Control
Number analyzed (Participants) | 10 | 10 | 10
units on a scale
  Baseline | 49 [43.88 to 73] | 53.75 [48.62 to 63] | 49.25 [41 to 57.5]
  After Treatment | 26.5 [16.87 to 39.75] | 50.25 [42 to 58.37] | 46.25 [37.5 to 54.12]
  4 weeks After Treatment | 29.25 [16.37 to 29.25] | 47.5 [41.37 to 61.37] | 44.5 [38.87 to 53.62]
Statistical Analysis 1: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of baseline values; Test type: Superiority; p = 0.643, Kruskal-Wallis
Statistical Analysis 2: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.018, Kruskal-Wallis
Statistical Analysis 3: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.027, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Kinesiotaping vs Sham Taping; Comparison of baseline values; Test type: Superiority; p = 0.677, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 5: Comparison: Kinesiotaping vs Control; Comparison of baseline values; Test type: Superiority; p = 0.677, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 6: Comparison: Sham Taping vs Control; Comparison of baseline values; Test type: Superiority; p = 0.326, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 7: Comparison: Kinesiotaping vs Sham Taping; Comparison of After Treatment Values; Test type: Superiority; p = 0.019, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 8: Comparison: Kinesiotaping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.014, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 9: Comparison: Sham Taping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.427, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 10: Comparison: Kinesiotaping vs Sham Taping; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.023, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 11: Comparison: Kinesiotaping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.021, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 12: Comparison: Sham Taping vs Control; Comparison of 4 week After Treatment Value; Test type: Superiority; p = 0.545, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 13: Comparison: Kinesiotaping; Test type: Superiority; p = 0.004, Friedman's two-way analysis of variance
Statistical Analysis 14: Comparison: Sham Taping; Test type: Superiority; p = 0.670, Friedman's two-way analysis of variance
Statistical Analysis 15: Comparison: Control; Test type: Superiority; p = 0.192, Friedman's two-way analysis of variance

2. Secondary Outcome: The Disabilities of the Arm, Shoulder and Hand Score (QuickDash)
Description: The patients will be requested to score from 1 to 5 points any difficulty experienced during different daily activities related to the upper extremity. Test has 1 module of compulsory items and two optional modules: work module (4 items) and sport/performing arts module (4 items). Scores range from 0 to 100, where higher scores indicate more disability.
Time Frame: 0. week (Baseline), 2. week (After Treatment), 6. week (4 weeks After Treatment)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Kinesiotaping | Sham Taping | Control
Number analyzed (Participants) | 10 | 10 | 10
score on a scale
  Baseline | 50 [41.5 to 74.43] | 46.57 [38.6 to 62.49] | 46.59 [33.81 to 57.39]
  After Treatment | 29.5 [10.4 to 59.7] | 47.72 [38.04 to 53.97] | 39.77 [33.52 to 49.42]
  4 weeks After Treatmentt | 18.18 [4.55 to 34.1] | 47.72 [34.62 to 56.81] | 39.75 [31.81 to 46.59]
Statistical Analysis 1: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of Before Treatment Values; Test type: Superiority; p = 0.633, Kruskal-Wallis
Statistical Analysis 2: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.282, Kruskal-Wallis
Statistical Analysis 3: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.015, Kruskal-Wallis
Statistical Analysis 4: Comparison: Kinesiotaping vs Sham Taping; Comparison of Before Treatment Values; Test type: Superiority; p = 0.677, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 5: Comparison: Kinesiotaping vs Control; Comparison of Before Treatment Values; Test type: Superiority; p = 0.344, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 6: Comparison: Sham Taping vs Control; Comparison of Before Treatment Values; Test type: Superiority; p = 0.596, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 7: Comparison: Kinesiotaping vs Sham Taping; Comparison of After Treatment Values; Test type: Superiority; p = 0.161, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 8: Comparison: Kinesiotaping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.257, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 9: Comparison: Sham Taping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.449, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 10: Comparison: Kinesiotaping vs Sham Taping; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.013, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 11: Comparison: Kinesiotaping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.019, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 12: Comparison: Sham Taping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.325, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 13: Comparison: Kinesiotaping; Test type: Superiority; p = 0.003, Friedman's two-way analysis of variance
Statistical Analysis 14: Comparison: Sham Taping; Test type: Superiority; p = 0.323, Friedman's two-way analysis of variance
Statistical Analysis 15: Comparison: Control; Test type: Superiority; p = 0.641, Friedman's two-way analysis of variance

3. Secondary Outcome: Visual Analogue Scale (VAS) at Rest
Description: Pain on lateral epicondyle at rest during the day was evaluated with the visual analog scale (VAS 0-10 cm). Higher score indicates more pain.
Time Frame: 0. week (Baseline), Immediate Effect (right after first taping in KT and sham taping groups), 2. week (After Treatment) and 6. week (4 weeks After Treatment)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Kinesiotaping | Sham Taping | Control
Number analyzed (Participants) | 10 | 10 | 10
score on a scale
  Baseline | 1.5 [0 to 3.25] | 1.5 [0 to 3.25] | 3 [0 to 4]
  Immediate Effect | 0 [0 to 0.5] | 1.5 [0 to 3.25] | NA [NA to NA] — Immediate effect assessments of tapings are not applicable to control group.
  After Treatment | 0 [0 to 0.25] | 0.5 [0 to 3] | 1 [0 to 3.5]
  4 weeks After Treatment | 0 [0 to 0] | 1 [0 to 3.25] | 1.5 [0.75 to 3]
Statistical Analysis 1: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of Baseline Values; Test type: Superiority; p = 0.715, Kruskal-Wallis
Statistical Analysis 2: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.227, Kruskal-Wallis
Statistical Analysis 3: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.012, Kruskal-Wallis
Statistical Analysis 4: Comparison: Kinesiotaping vs Sham Taping; Comparison of Baseline Values; Test type: Superiority; p = 0.907, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 5: Comparison: Kinesiotaping vs Control; Comparison of Baseline Values; Test type: Superiority; p = 0.482, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 6: Comparison: Kinesiotaping vs Control; Comparison of Baseline Values; Test type: Superiority; p = 0.485, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 7: Comparison: Kinesiotaping vs Sham Taping; Comparison of After Treatment Values; Test type: Superiority; p = 0.129, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 8: Comparison: Kinesiotaping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 9: Comparison: Sham Taping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.935, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 10: Comparison: Kinesiotaping vs Sham Taping; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 11: Comparison: Kinesiotaping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.036, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 12: Comparison: Sham Taping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.056, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 13: Comparison: Kinesiotaping; Test type: Superiority; p = 0.016, Friedman's two-way analysis of variance
Statistical Analysis 14: Comparison: Sham Taping; Test type: Superiority; p = 0.618, Friedman's two-way analysis of variance
Statistical Analysis 15: Comparison: Control; Test type: Superiority; p = 0.48, Friedman's two-way analysis of variance
Statistical Analysis 16: Comparison: Kinesiotaping vs Sham Taping; Comparison of immediate effect between groups; Test type: Superiority; p = 0.034, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Kinesiotaping; Immediate effect compared to baseline; Test type: Superiority; p = 0.041, Kruskal-Wallis
Statistical Analysis 18: Comparison: Sham Taping; Immediate effect compared to baseline; Test type: Superiority; p = 1, Kruskal-Wallis

4. Secondary Outcome: Visual Analogue Scale (VAS) at Daily Activity
Description: Pain on lateral epicondyle during daily activity was evaluated with the visual analog scale (VAS 0-10 cm). Higher score indicates more pain.
Time Frame: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Kinesiotaping | Sham Taping | Control
Number analyzed (Participants) | 10 | 10 | 10
score on a scale
  Baseline | 6.5 [5 to 7.25] | 7.5 [6.75 to 8] | 7 [5 to 7]
  Immediate Effect | 5 [1.5 to 6.25] | 7 [6 to 8] | NA [NA to NA] — Immediate effect assessments of tapings are not applicable to control group.
  After Treatment | 3 [2 to 5] | 7 [5.75 to 8] | 5 [5 to 7]
  4 weeks After Treatment | 3 [1.75 to 5.25] | 6.5 [4.75 to 7.25] | 5.5 [5 to 7]
Statistical Analysis 1: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of Baseline Values; Test type: Superiority; p = 0.103, Kruskal-Wallis
Statistical Analysis 2: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.002, Kruskal-Wallis
Statistical Analysis 3: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.008, Kruskal-Wallis
Statistical Analysis 4: Comparison: Kinesiotaping vs Sham Taping; Comparison of Baseline Values; Test type: Superiority; p = 0.76, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 5: Comparison: Kinesiotaping vs Control; Comparison of Baseline Values; Test type: Superiority; p = 1, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 6: Comparison: Sham Taping vs Control; Comparison of Baseline Values; Test type: Superiority; p = 0.056, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 7: Comparison: Kinesiotaping vs Sham Taping; Comparison of After Treatment Values; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 8: Comparison: Kinesiotaping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 9: Comparison: Sham Taping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.117, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 10: Comparison: Kinesiotaping vs Sham Taping; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.006, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 11: Comparison: Kinesiotaping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.013, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 12: Comparison: Sham Taping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.487, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 13: Comparison: Kinesiotaping; Test type: Superiority; p = 0.002, Friedman's two-way analysis of variance
Statistical Analysis 14: Comparison: Sham Taping; Test type: Superiority; p = 0.102, Friedman's two-way analysis of variance
Statistical Analysis 15: Comparison: Control; Test type: Superiority; p = 0.165, Friedman's two-way analysis of variance
Statistical Analysis 16: Comparison: Kinesiotaping vs Sham Taping; Comparison of immediate effect between groups; Test type: Superiority; p = 0.007, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Kinesiotaping; Immediate effect compared to baseline; Test type: Superiority; p = 0.028, Kruskal-Wallis
Statistical Analysis 18: Comparison: Sham Taping; Immediate effect compared to baseline; Test type: Superiority; p = 0.83, Kruskal-Wallis

5. Secondary Outcome: Visual Analogue Scale (VAS) at Night
Description: Pain on lateral epicondyle at night was evaluated with the visual analog scale (VAS 0-10 cm). Higher score indicates more pain.
Time Frame: 0. week (Baseline), 2. week (After Treatment), 6. week (4 weeks After Treatment)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Kinesiotaping | Sham Taping | Control
Number analyzed (Participants) | 10 | 10 | 10
score on a scale
  Before Treatment | 2.5 [0 to 4.5] | 2.5 [0 to 3.5] | 3.5 [0 to 5.75]
  After Treatment | 0 [0 to 0.25] | 2 [0 to 3.5] | 1 [0 to 3.25]
  4 weeks After Treatment | 0 [0 to 0] | 2 [0 to 3.25] | 0 [0 to 3.25]
Statistical Analysis 1: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of Baseline Values; Test type: Superiority; p = 0.837, Kruskal-Wallis
Statistical Analysis 2: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.215, Kruskal-Wallis
Statistical Analysis 3: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.078, Kruskal-Wallis
Statistical Analysis 4: Comparison: Kinesiotaping vs Sham Taping; Comparison of Baseline Values; Test type: Superiority; p = 0.699, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 5: Comparison: Kinesiotaping vs Control; Comparison of Baseline Values; Test type: Superiority; p = 0.846, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 6: Comparison: Sham Taping vs Control; Comparison of Baseline Values; Test type: Superiority; p = 0.56, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 7: Comparison: Kinesiotaping vs Sham Taping; Comparison of After Treatment Values; Test type: Superiority; p = 0.087, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 8: Comparison: Kinesiotaping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.183, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 9: Comparison: Sham Taping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.719, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 10: Comparison: Kinesiotaping vs Sham Taping; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.023, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 11: Comparison: Kinesiotaping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.196, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 12: Comparison: Sham Taping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.318, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 13: Comparison: Kinesiotaping; Test type: Superiority; p = 0.001, Friedman's two-way analysis of variance
Statistical Analysis 14: Comparison: Sham Taping; Test type: Superiority; p = 0.483, Friedman's two-way analysis of variance
Statistical Analysis 15: Comparison: Control; Test type: Superiority; p = 0.004, Friedman's two-way analysis of variance

6. Secondary Outcome: Painless Grip Strength
Description: Grip strength will be measured using a hand held dynamometer (JAMAR, Sammons Preston, Inc., Bolingbrook, IL). Patients will be asked to grip the dynamometer until (s)he feel pain in elbow. Three evaluations will be made with resting periods in between and average scores will be recorded.
Time Frame: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Kinesiotaping | Sham Taping | Control
Number analyzed (Participants) | 10 | 10 | 10
kg
  Baseline | 14 [8 to 19.75] | 12 [2 to 25] | 13 [9.5 to 20.5]
  Immediate Effect | 17 [10 to 23] | 13 [3.75 to 27.75] | NA [NA to NA] — Immediate effect assessments of tapings are not applicable to control group.
  After Treatment | 17.5 [14.75 to 28.25] | 13 [10 to 21.25] | 15 [9.5 to 20.5]
  4 weeks After Treatment | 20 [17 to 28.75] | 14.5 [10 to 24.5] | 14.5 [9.5 to 20.5]
Statistical Analysis 1: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of Baseline Values; Test type: Superiority; p = 0.897, Kruskal-Wallis
Statistical Analysis 2: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.325, Kruskal-Wallis
Statistical Analysis 3: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.172, Kruskal-Wallis
Statistical Analysis 4: Comparison: Kinesiotaping vs Sham Taping; Comparison of Baseline Values; Test type: Superiority; p = 0.622, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 5: Comparison: Kinesiotaping vs Control; Comparison of Baseline Values; Test type: Superiority; p = 0.909, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 6: Comparison: Sham Taping vs Control; Comparison of Baseline Values; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 7: Comparison: Kinesiotaping vs Sham Taping; Comparison of After Treatment Values; Test type: Superiority; p = 0.24, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 8: Comparison: Kinesiotaping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.161, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 9: Comparison: Sham Taping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.909, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 10: Comparison: Kinesiotaping vs Sham Taping; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.255, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 11: Comparison: Kinesiotaping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.058, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 12: Comparison: Sham Taping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.569, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 13: Comparison: Kinesiotaping; Test type: Superiority; p = 0.007, Friedman's two-way analysis of variance
Statistical Analysis 14: Comparison: Sham Taping; Test type: Superiority; p = 0.614, Friedman's two-way analysis of variance
Statistical Analysis 15: Comparison: Control; Test type: Superiority; p = 0.072, Friedman's two-way analysis of variance
Statistical Analysis 16: Comparison: Kinesiotaping vs Sham Taping; Comparison of immediate effect between groups; Test type: Superiority; p = 0.447, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Kinesiotaping; Immediate effect compared to baseline; Test type: Superiority; p = 0.084, Kruskal-Wallis
Statistical Analysis 18: Comparison: Sham Taping; Immediate effect compared to baseline; Test type: Superiority; p = 0.235, Kruskal-Wallis

7. Secondary Outcome: Grip Strength
Description: Grip strength will be measured using a hand held dynamometer (JAMAR, Sammons Preston, Inc., Bolingbrook, IL). Patients will be asked to grip with maximum strength. Three evaluations will be made with resting periods in between and average scores will be recorded.
Time Frame: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Kinesiotaping | Sham Taping | Control
Number analyzed (Participants) | 10 | 10 | 10
kg
  Baseline | 20 [14.75 to 27.5] | 19.5 [14.75 to 30.25] | 23.5 [15 to 28.25]
  Immediate Effect | 22 [16.5 to 29.25] | 19.5 [14.5 to 32.5] | NA [NA to NA] — Immediate effect assessments of tapings are not applicable to control group.
  After Treatment | 22.5 [17.5 to 29.25] | 20 [14.5 to 27.25] | 24 [19 to 25.75]
  4 weeks After Treatment | 25 [21.5 to 28.75] | 21 [12 to 28] | 24 [18.5 to 27]
Statistical Analysis 1: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of Baseline Values; Test type: Superiority; p = 0.958, Kruskal-Wallis
Statistical Analysis 2: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.597, Kruskal-Wallis
Statistical Analysis 3: Comparison: Kinesiotaping vs Sham Taping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.518, Kruskal-Wallis
Statistical Analysis 4: Comparison: Kinesiotaping vs Sham Taping; Comparison of Baseline Values; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 5: Comparison: Kinesiotaping vs Control; Comparison of Baseline Values; Test type: Superiority; p = 0.733, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 6: Comparison: Sham Taping vs Control; Comparison of Baseline Values; Test type: Superiority; p = 1, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 7: Comparison: Kinesiotaping vs Sham Taping; Comparison of After Treatment Values; Test type: Superiority; p = 0.404, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 8: Comparison: Kinesiotaping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.97, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 9: Comparison: Sham Taping vs Control; Comparison of After Treatment Values; Test type: Superiority; p = 0.362, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 10: Comparison: Kinesiotaping vs Sham Taping; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.271, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 11: Comparison: Kinesiotaping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.519, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 12: Comparison: Sham Taping vs Control; Comparison of 4 week After Treatment Values; Test type: Superiority; p = 0.569, Wilcoxon (Mann-Whitney) — p-value is adjusted for multiple comparisons; p<0.017 is significant
Statistical Analysis 13: Comparison: Kinesiotaping; Test type: Superiority; p = 0.004, Friedman's two-way analysis of variance
Statistical Analysis 14: Comparison: Sham Taping; Test type: Superiority; p = 0.973, Friedman's two-way analysis of variance
Statistical Analysis 15: Comparison: Control; Test type: Superiority; p = 0.886, Friedman's two-way analysis of variance
Statistical Analysis 16: Comparison: Kinesiotaping vs Sham Taping; Comparison of immediate effect between groups; Test type: Superiority; p = 0.82, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Kinesiotaping; Immediate effect compared to baseline; Test type: Superiority; p = 0.017, Kruskal-Wallis
Statistical Analysis 18: Comparison: Sham Taping; Immediate effect compared to baseline; Test type: Superiority; p = 0.734, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Kinesiotaping: Kinesio taping by using space correction and fascia correction techniques every 3 days for 2 weeks in addition to exercises
  Kinesio taping: Kinesio tape will be applied by using space correction and fascia correction technique on forearm of the patients for the treatment of lateral epicondylitis
  Exercise: Stretching exercises of wrist 30 seconds to one minute, twice a day and strengthening exercises will performed be 10 repetitions in 2 or 3 series.
  No adverse effect occured.
- Sham Taping: Sham taping without using any techniques every 3 days for 2 weeks in addition to exercises
  Sham taping: Sham taping will be performed without using any technique
  Exercise: Stretching exercises of wrist 30 seconds to one minute, twice a day and strengthening exercises will performed be 10 repetitions in 2 or 3 series.
  No adverse effect occured.
- Control: Stretching and strengthening exercises of wrist
  Exercise: Stretching exercises of wrist 30 seconds to one minute, twice a day and strengthening exercises will performed be 10 repetitions in 2 or 3 series.
  No adverse effect occured.
Arm/Group | Kinesiotaping | Sham Taping | Control
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 1/11 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kinesiotaping (N=11) | Sham Taping (N=11) | Control (N=11)
Allergy to Tape (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Contact dermatitis due to tape

LIMITATIONS AND CAVEATS:
The limitations of this study are small sample size and relatively short follow-up time. Also, only patients with symptom duration less than 12 weeks were included so results of the study can not be generalized for chronic lateral epicondylitis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03074500/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03074500/SAP_001.pdf